CLINICAL TRIAL: NCT01139762
Title: A Phase 3b, Randomized, Double-blind, Placebo-controlled Parallel-design Study to Evaluate the Efficacy and Safety of Tadalafil Co-administered With Finasteride for 6 Months in Men With Lower Urinary Tract Symptoms and Prostatic Enlargement Secondary to Benign Prostatic Hyperplasia
Brief Title: A Study of Tadalafil Use With Finasteride in Men With Enlarged Prostates and Urinary Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13529; H6D-CR-LVIW (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-06-01; First posted 2010-06-09 (Estimated); Results first posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-01

CONDITIONS: Benign Prostatic Hyperplasia; Enlarged Prostate
Keywords: Benign Prostatic Hyperplasia (BPH); Enlarged Prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil; Finasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil (Experimental)
  Interventions: Drug: Tadalafil; Drug: Finasteride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Finasteride

INTERVENTIONS:
Drug: Tadalafil — 5 milligrams (mg) administered orally, once daily for 26 weeks
  Other Names: Cialis; LY#450190
  Arms: Tadalafil
Drug: Placebo — Administered orally, once daily for 26 weeks
  Arms: Placebo
Drug: Finasteride — 5mg administered orally, once daily for 26 weeks

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of once daily tadalafil when taken with finasteride as a treatment for men with signs and symptoms of Benign Prostatic Hyperplasia and demonstrable prostate enlargement.

ELIGIBILITY:
Inclusion Criteria:

* Have not taken the following treatments within the indicated duration and agree not to use at any time during the study:

  * All other Benign Prostatic Hyperplasia (BPH) therapy (including herbal preparations) for at least 4 weeks prior to receiving study medication.
  * Overactive bladder therapy (including antimuscarinics) for at least 4 weeks prior to receiving study medication.
  * Erectile Dysfunction therapy (including herbal preparations) for at least 4 weeks prior to receiving study medication.
  * Finasteride or dutasteride use at any time.
* Have bladder outlet obstruction as defined by a urinary peak flow rate (Qmax) of greater than or equal to 4 and less than or equal to 15 milliliters (mL)/second before receiving study drug.
* Have prostate enlargement measured by ultrasound at screening.

Exclusion Criteria:

* Have prostate cancer, are being treated for cancer or have clinical evidence of prostate cancer [Prostate-specific antigen (PSA) greater than 10 nanograms/milliliter (ng/mL) at the start of study].
* Have had any of the following in the past 90 days: Heart attack, also known as a myocardial infarction (MI); Heart bypass surgery (called coronary artery bypass graft surgery); Had a procedure to open up blood vessels in the heart known as angioplasty or stent placement (percutaneous coronary intervention).
* Have problems with kidneys, liver, or nervous system
* Have uncontrolled diabetes
* Have had a stroke or a significant injury to brain or spinal cord.
* Have scheduled or planned surgery during the course of the study.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (65):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Davis, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laguna Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vacaville, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sarasota, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Georgetown, Texas
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edegem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kortrijk
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Abbottsford, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Surrey, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitchener, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North York, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thunder Bay, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pointe-Claire, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trois-Rivières, Quebec
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suresnes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vandœuvre-lès-Nancy
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hettstedt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mühlacker
- Greece (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Larissa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sassari
- Mexico (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saltillo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tlalpan
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kutno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zabrze
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
- Turkey (Türkiye) (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denizli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir

REFERENCES:
- [Derived] Glina S, Roehrborn CG, Esen A, Plekhanov A, Sorsaburu S, Henneges C, Buttner H, Viktrup L. Sexual function in men with lower urinary tract symptoms and prostatic enlargement secondary to benign prostatic hyperplasia: results of a 6-month, randomized, double-blind, placebo-controlled study of tadalafil coadministered with finasteride. J Sex Med. 2015 Jan;12(1):129-38. doi: 10.1111/jsm.12714. Epub 2014 Oct 29. PMID 25353053

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 3 periods: a 4-week washout period, a 4-week, single-blind, placebo lead-in period, and a 26-week double-blind randomized active treatment period. Participants who did not complete the washout and placebo lead-in period were considered screen failures.
Groups:
- Screening-Washout and Placebo Lead-In: 4 weeks washout period and followed by placebo orally, once daily for 4 weeks during placebo lead-in period.
- Tadalafil: 5 milligrams (mg) Tadalafil orally, once daily co-administered with 5 mg Finasteride orally, once daily for 26 weeks during double-blind randomized active treatment period.
- Placebo: Placebo orally, once daily co-administered with 5 mg Finasteride orally, once daily for 26 weeks during double-blind randomized active treatment period.
Period: Washout and Placebo Lead-In Period
Arm/Group | Screening-Washout and Placebo Lead-In | Tadalafil | Placebo
Started | 1070 | 0 | 0
Completed | 696 | 0 | 0
Not Completed | 374 | 0 | 0
Not completed — Entry Criteria Not Met | 258 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 83 | 0 | 0
Not completed — Physician Decision | 12 | 0 | 0
Not completed — Sponsor Decision | 10 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0
Period: Double-Blind Randomized Active Treatment
Arm/Group | Screening-Washout and Placebo Lead-In | Tadalafil | Placebo
Started | 0 | 346 | 350
Received at Least 1 Dose of Study Drug | 0 | 345 | 350
Completed | 0 | 306 | 286
Not Completed | 0 | 40 | 64
Not completed — Adverse Event | 0 | 4 | 10
Not completed — Death | 0 | 1 | 1
Not completed — Entry Criteria Not Met | 0 | 14 | 17
Not completed — Protocol Violation | 0 | 2 | 8
Not completed — Withdrawal by Subject | 0 | 6 | 13
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Sponsor Decision | 0 | 5 | 6
Not completed — Lack of Efficacy | 0 | 3 | 5
Not completed — Lost to Follow-up | 0 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Tadalafil: 5 milligrams (mg) Tadalafil orally, once daily co-administered with 5 mg Finasteride orally, once daily for 26 weeks.
- Placebo: Placebo orally, once daily co-administered with 5 mg Finasteride orally, once daily for 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Tadalafil | Placebo | Total
Number analyzed (Participants) | 345 | 350 | 695
Age Continuous [Mean (Standard Deviation); unit: years] | 63.8 (7.50) | 63.6 (7.85) | 63.7 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 345 | 350 | 695
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Information was not collected for participants outside of United States.
  Participants
    Hispanic or Latino | 4 | 5 | 9
    Not Hispanic or Latino | 39 | 41 | 80
    Unknown or Not Reported | 302 | 304 | 606
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 33 | 37 | 70
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 15 | 21
  White | 298 | 296 | 594
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 46 | 89
  Greece | 18 | 12 | 30
  Turkey | 26 | 19 | 45
  Russian Federation | 32 | 37 | 69
  Italy | 21 | 25 | 46
  France | 21 | 9 | 30
  Mexico | 33 | 37 | 70
  Canada | 30 | 28 | 58
  Argentina | 46 | 41 | 87
  Belgium | 7 | 16 | 23
  Poland | 32 | 39 | 71
  Brazil | 12 | 13 | 25
  Germany | 24 | 28 | 52
Lower urinary tract symptoms (LUTS) severity [Number; unit: participants] — The International Prostate Symptom Score (IPSS) is a rating scale for severity of lower urinary tract symptoms (LUTS). The IPSS has a 7-component questionnaire. Each question is scored on a scale from 0 (none/no symptoms) to 5 (frequent symptoms), for a total score range of 0 to 35. Higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
  participants
    Moderate (IPSS<20) | 238 | 235 | 473
    Severe (IPSS≥20) | 106 | 114 | 220
    Unknown | 1 | 1 | 2
Peak urine flow rate [Number; unit: participants] — Peak urine flow rate is expressed as milliliters/second (mL/sec).
  participants
    <10 milliliters/second (mL/sec) | 154 | 169 | 323
    10-15 mL/sec | 190 | 180 | 370
    >15 mL/sec | 1 | 1 | 2
Postvoid residual volume (PVR) [Mean (Standard Deviation); unit: milliliters (mL)] — Two participants from placebo group had missing data and are not included in the calculation of mean and standard deviation.
  milliliters (mL) | 65.5 (60.69) | 62.6 (59.57) | 64.1 (60.10)
Prostate Volume [Mean (Standard Deviation); unit: milliliters (mL)] | 48.2 (19.43) | 50.6 (21.17) | 49.4 (20.35)
Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)] — One participant from Tadalafil and 3 participants from placebo group had missing data and are not included in the calculation of mean and standard deviation.
  nanograms/milliliter (ng/mL) | 2.3 (2.02) | 2.5 (2.06) | 2.4 (2.04)
Erectile Dysfunction [Number; unit: participants]
  Yes | 227 | 223 | 450
  No | 118 | 127 | 245
Sexual activity with female partner [Number; unit: participants]
  Yes | 305 | 305 | 610
  No | 40 | 44 | 84
  Not Applicable | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 173.5 (7.90) | 173.8 (7.65) | 173.7 (7.77)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 85.3 (14.16) | 85.6 (14.16) | 85.4 (14.15)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meter (kg/m²)] | 28.3 (4.00) | 28.3 (3.80) | 28.3 (3.90)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total International Prostate Symptom Score (IPSS) From Baseline to 12 Weeks
Description: The International Prostate Symptom Score (IPSS) is a rating scale for severity of lower urinary tract symptoms (LUTS). The IPSS has a 7-component questionnaire. Each question is scored on a scale from 0 (none/no symptoms) to 5 (frequent symptoms), for a total score range of 0 to 35. Higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Least Squares (LS) Mean values were obtained from a mixed model repeated measures (MMRM) analysis. Model includes treatment, region, visit, baseline total IPSS, and visit-by-treatment interaction.
Time Frame: Baseline, 12 weeks
Population: All randomized participants who received at least 1 dose of the study drug, had baseline and at least 1 post-baseline IPSS measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 345 | 350
units on a scale | -5.18 (0.32) | -3.76 (0.32)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; MMRM model includes treatment, region, visit, and treatment-by-visit interaction as fixed effects, and subject as a random effect. Baseline total IPSS was the covariate. No imputation of missing total IPSS data was performed. The within-subject errors were modeled using an unstructured covariance structure; Test type: Superiority or Other; p = 0.001, Mixed Model Repeated Measures Analysis; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = -1.41, 95% CI 2-sided [-2.27 to -0.55]

2. Secondary Outcome: Change in Total International Prostate Symptom Score (IPSS) From Baseline to 4 and 26 Weeks
Description: as for outcome 1
Time Frame: Baseline, 4 weeks, 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 345 | 350
units on a scale
  4 weeks | -3.95 (0.29) | -2.29 (0.28)
  26 weeks | -5.51 (0.33) | -4.47 (0.33)

3. Secondary Outcome: Change in International Prostate Symptom Score (IPSS) Subscores Index From Baseline to 4, 12, and 26 Weeks
Description: IPSS storage (irritative) subscore is the sum of Questions 2, 4 and 7 of the 7-component IPSS questionnaire. Scores range from 0 (no irritative symptoms) to 5 (frequent irritative symptoms), with total subscore of the 3 questions for irritative subscore range from 0 to 15. IPSS voiding (obstructive) subscore is the sum of Questions 1, 3, 5 and 6 of the IPSS questionnaire. Scores range from 0 (no obstructive symptoms) to 5 (frequent obstructive symptoms), with total subscore of the 4 questions of the obstructive score range from 0 to 20. Least Squares (LS) Mean values were obtained from a mixed model repeated measures (MMRM) analysis. Model includes treatment, region, visit, baseline total IPSS, and visit-by-treatment interaction.
Time Frame: Baseline, 4 weeks, 12 weeks, 26 weeks
Population: All randomized participants who received at least 1 dose of the study drug, had baseline and at least 1 post-baseline IPSS subscore measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 345 | 350
units on a scale
  IPSS storage (irritative) subscore - 4 weeks | -1.27 (0.14) | -0.76 (0.14)
  IPSS storage (irritative) subscore - 12 weeks | -1.74 (0.14) | -1.34 (0.14)
  IPSS storage (irritative) subscore - 26 weeks | -2.00 (0.15) | -1.66 (0.15)
  IPSS voiding (obstructive) subscore - 4 weeks | -2.65 (0.19) | -1.47 (0.19)
  IPSS voiding (obstructive) subscore - 12 weeks | -3.41 (0.21) | -2.37 (0.21)
  IPSS voiding (obstructive) subscore - 26 weeks | -3.50 (0.22) | -2.77 (0.22)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.007, Mixed Model Repeated Measures Analysis — P-value is for IPSS storage (irritative) subscore - 4 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = -0.51, 95% CI 2-sided [-0.87 to -0.14]
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.040, Mixed Model Repeated Measures Analysis — P-value is for IPSS storage (irritative) subscore - 12 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = -0.41, 95% CI 2-sided [-0.80 to -0.02]
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.107, Mixed Model Repeated Measures Analysis — P-value is for IPSS storage (irritative) subscore - 26 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = -0.34, 95% CI 2-sided [-0.75 to 0.07]
Statistical Analysis 4: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for IPSS voiding (obstructive) subscore - 4 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = -1.18, 95% CI 2-sided [-1.69 to -0.68]
Statistical Analysis 5: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for IPSS voiding (obstructive) subscore - 12 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = -1.04, 95% CI 2-sided [-1.62 to -0.46]
Statistical Analysis 6: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.015, Mixed Model Repeated Measures Analysis — P-value is IPSS voiding (obstructive) subscore - 26 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = -0.73, 95% CI 2-sided [-1.32 to -0.14]

4. Secondary Outcome: Change in International Prostate Symptom Score (IPSS) Quality of Life Index From Baseline to 4, 12, and 26 Weeks
Description: IPSS Quality of Life Index assesses participant response to the following question: "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?" Response options are Delighted (0); Pleased (1); Mostly satisfied (2); Mixed-about equally satisfied and dissatisfied (3); Mostly dissatisfied (4); Unhappy (5); Terrible (6), with a total range of 0-6. Least Squares (LS) Mean values were obtained from a mixed model repeated measures (MMRM) analysis. Model includes treatment, region, visit, baseline total IPSS, and visit-by-treatment interaction.
Time Frame: Baseline, 4 weeks, 12 weeks, 26 weeks
Population: All randomized participants who received at least 1 dose of the study drug, had baseline and at least 1 post-baseline IPSS quality of life measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 345 | 350
units on a scale
  4 weeks | -0.63 (0.07) | -0.32 (0.06)
  12 weeks | -0.95 (0.07) | -0.76 (0.07)
  26 weeks | -1.10 (0.08) | -0.92 (0.08)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 4 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = -0.32, 95% CI 2-sided [-0.50 to -0.14]
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.051, Mixed Model Repeated Measures Analysis — P-value is for 12 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = -0.19, 95% CI 2-sided [-0.38 to 0.00]
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.107, Mixed Model Repeated Measures Analysis — P-value is for 26 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = -0.17, 95% CI 2-sided [-0.38 to 0.04]

5. Secondary Outcome: Change in International Index of Erectile Function (IIEF) - Erectile Function Domain Scores From Baseline to 4, 12, and 26 Weeks
Description: Self-reported erectile function over the past 4 weeks. IIEF- EF is the sum of Questions 1-5 and 15 of the IIEF. Questions 1-5 are scored 0 (low/no erectile function) to 5 (high erectile function) and Question 15 is scored 1 (very low confidence) to 5 (very high confidence), for a total score ranging from 1 to 30. Higher scores represent better erectile function. Least Squares (LS) Mean values were obtained from a mixed model repeated measures (MMRM) analysis. Model includes treatment, region, visit, baseline IIEF, and visit-by-treatment interaction.
Time Frame: Baseline, 4 weeks, 12 weeks, 26 weeks
Population: All randomized participants who were sexually active with female partner and had erectile dysfunction (ED), received at least 1 dose of the study drug, had baseline and at least 1 post-baseline IIEF-EF measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 203 | 201
units on a scale
  4 weeks | 3.71 (0.50) | -1.14 (0.51)
  12 weeks | 4.71 (0.56) | 0.63 (0.57)
  26 weeks | 4.71 (0.57) | -0.02 (0.60)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; MMRM model includes treatment, region, visit, and treatment-by-visit interaction as fixed effects, and subject as a random effect. Baseline IIEF was the covariate. No imputation of missing IIEF data was performed. The within-subject errors were modeled using an unstructured covariance structure; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 4 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 4.85, 95% CI 2-sided [3.49 to 6.21]
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 12 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 4.08, 95% CI 2-sided [2.55 to 5.60]
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 26 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 4.73, 95% CI 2-sided [3.15 to 6.31]

6. Secondary Outcome: Change in International Index of Erectile Function (IIEF) - Overall Satisfaction Domain Scores From Baseline to 4, 12, and 26 Weeks
Description: Self-reported overall satisfaction over the past 4 weeks. IIEF-Overall Satisfaction is the sum of Questions 13 and 14 of IIEF questionnaire. Scores range from 1 (low/no satisfaction) to 5 (high satisfaction) for each question, with the total possible score for the 2 questions ranging from 2 to 10. Higher total scores indicate higher satisfaction. Least Squares (LS) Mean values were obtained from a mixed model repeated measures (MMRM) analysis. Model includes treatment, region, visit, baseline IIEF, and visit-by-treatment interaction.
Time Frame: Baseline, 4 weeks, 12 weeks, 26 weeks
Population: All randomized participants who were sexually active with female partner and had erectile dysfunction (ED), received at least 1 dose of the study drug, had baseline and at least 1 post-baseline IIEF-Overall Satisfaction measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 203 | 201
units on a scale
  4 weeks | 0.91 (0.15) | -0.10 (0.15)
  12 weeks | 1.38 (0.16) | 0.31 (0.17)
  26 weeks | 1.61 (0.17) | 0.40 (0.18)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 4 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 1.01, 95% CI 2-sided [0.61 to 1.40]
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 12 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 1.06, 95% CI 2-sided [0.61 to 1.51]
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 26 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 1.22, 95% CI 2-sided [0.74 to 1.69]

7. Secondary Outcome: Change in International Index of Erectile Function (IIEF) - Intercourse Satisfaction Domain Scores From Baseline to 4, 12, and 26 Weeks
Description: Self-reported intercourse satisfaction over the past 4 weeks. IIEF-intercourse satisfaction is the sum of Questions 6, 7 and 8 of the IIEF. Scores range from 0 (low/no satisfaction) to 5 (high satisfaction) for each question, with the total possible score for the 3 questions of 0 to 15. Higher total scores indicate higher satisfaction. Least Squares (LS) Mean values were obtained from a mixed model repeated measures (MMRM) analysis. Model includes treatment, region, visit, baseline IIEF, and visit-by-treatment interaction.
Time Frame: Baseline, 4 weeks, 12 weeks, 26 weeks
Population: All randomized participants who were sexually active with female partner and had erectile dysfunction (ED), received at least 1 dose of the study drug, had baseline and at least 1 post-baseline IIEF-intercourse satisfaction measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 203 | 201
units on a scale
  4 weeks | 1.36 (0.24) | -0.46 (0.24)
  12 weeks | 1.68 (0.26) | 0.08 (0.27)
  26 weeks | 1.72 (0.27) | -0.26 (0.28)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 4 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 1.82, 95% CI 2-sided [1.18 to 2.47]
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 12 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 1.59, 95% CI 2-sided [0.88 to 2.31]
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 26 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 1.98, 95% CI 2-sided [1.23 to 2.73]

8. Secondary Outcome: Change in International Index of Erectile Function (IIEF) - Orgasmic Function Domain Scores From Baseline to 4, 12, and 26 Weeks
Description: Orgasmic Function domain scores is the sum of Questions 9 and 10 from the IIEF questionnaire. Scores range from 0 (low/no orgasm) to 5 (high orgasm) for each question, with the total possible score for the 2 questions ranging from 0 to 10. Higher total scores indicate higher orgasm. Least Squares (LS) Mean values were obtained from a mixed model repeated measures (MMRM) analysis. Model includes treatment, region, visit, baseline IIEF, and visit-by-treatment interaction.
Time Frame: Baseline, 4 weeks, 12 weeks, 26 weeks
Population: All randomized participants who were sexually active with female partner and had erectile dysfunction (ED), received at least 1 dose of the study drug, had baseline and at least 1 post-baseline IIEF-orgasmic function domain score measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 203 | 201
units on a scale
  4 weeks | 0.90 (0.22) | -0.63 (0.23)
  12 weeks | 1.08 (0.23) | 0.18 (0.24)
  26 weeks | 0.89 (0.24) | -0.18 (0.25)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 4 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 1.53, 95% CI 2-sided [0.92 to 2.13]
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.006, Mixed Model Repeated Measures Analysis — P-value is for 12 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 0.90, 95% CI 2-sided [0.27 to 1.54]
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.002, Mixed Model Repeated Measures Analysis — P-value is for 26 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 1.07, 95% CI 2-sided [0.41 to 1.74]

9. Secondary Outcome: Change in International Index of Erectile Function (IIEF) - Sexual Desire Domain Scores From Baseline to 4, 12, and 26 Weeks
Description: Sexual desire domain scores is the sum of Questions 11 and 12 from the IIEF questionnaire. Scores range from 1 (low/no desire) to 5 (high desire) for each question, with the total possible score for the 2 questions ranging from 2 to 10. Higher total scores indicate higher desire. Least Squares (LS) Mean values were obtained from a mixed model repeated measures (MMRM) analysis. Model includes treatment, region, visit, baseline IIEF, and visit-by-treatment interaction.
Time Frame: Baseline, 4 weeks, 12 weeks, 26 weeks
Population: All randomized participants who were sexually active with female partner and had erectile dysfunction (ED), received at least 1 dose of the study drug, had baseline and at least 1 post-baseline IIEF-sexual desire domain score measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 203 | 201
units on a scale
  4 weeks | 0.46 (0.12) | -0.47 (0.12)
  12 weeks | 0.56 (0.13) | -0.23 (0.13)
  26 weeks | 0.71 (0.13) | -0.05 (0.14)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 4 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 0.93, 95% CI 2-sided [0.61 to 1.25]
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 12 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 0.79, 95% CI 2-sided [0.44 to 1.14]
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for 26 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 0.76, 95% CI 2-sided [0.39 to 1.13]

10. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) at 26 Weeks
Description: Patient Global Impression of Improvement (PGI-I) measures the participant's perception of improvement at the time of assessment compared with the start of treatment. Number of participants is reported by the categorized score ranging from 1 (very much better) to 7 (very much worse).
Time Frame: 26 weeks
Population: All randomized participants who received at least 1 dose of the study drug and had PGI-I measurement at 26 weeks endpoint.
Measure: Number; unit: participants
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 309 | 288
participants
  1 = Very much better | 21 | 29
  2 = Much better | 124 | 82
  3 = Little better | 102 | 112
  4 = No change | 49 | 52
  5 = A little worse | 10 | 5
  6 = Much worse | 2 | 7
  7 = Very much worse | 1 | 1
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.034, Cochran-Mantel-Haenszel — P-value is for overall distribution of responses; Adjusted for baseline lower urinary tract symptoms (LUTS) severity

11. Secondary Outcome: Treatment Satisfaction Scale - Benign Prostatic Hyperplasia (TSS-BPH) at 26 Weeks
Description: The TSS-BPH was a validated participant-rated instrument that measured participant satisfaction with treatment based on a 13-item questionnaire. It consists of 10 items on a Likert-like scale with scores ranging from 1 (higher satisfaction) to 5 (lower satisfaction), 1 item with score ranging from 0 (higher satisfaction) to 5 (lower satisfaction), and 2 yes/no questions. The mean score for each participant ranges from 0.9 (higher satisfaction) to 5.0 (lower satisfaction). Data presented are the average of mean scores for each treatment group.
Time Frame: 26 weeks
Population: All randomized participants who received at least 1 dose of the study drug and had TSS-BPH measurement at 26 weeks endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 303 | 293
units on a scale | 2.0 (0.63) | 2.1 (0.66)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.031, Van Elteren test; Van Elteren test was stratified by region

12. Secondary Outcome: Clinician Global Impression of Improvement (CGI-I) at 26 Weeks
Description: Clinician Global Impression of Improvement (CGI-I) measures clinician's perception of participant improvement at the time of assessment compared with the start of treatment. Number of participants is reported by the categorized score ranging from 1 (very much better) to 7 (very much worse).
Time Frame: 26 weeks
Population: All randomized participants who received at least 1 dose of the study drug and had CGI-I measurement at 26 weeks endpoint.
Measure: Number; unit: participants
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 307 | 290
participants
  1 = Very much improved | 23 | 22
  2 = Much improved | 129 | 97
  3 = Minimally improved | 98 | 106
  4 = No change | 47 | 48
  5 = Minimally worse | 5 | 10
  6 = Much worse | 5 | 6
  7 = Very much worse | 0 | 1
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.328, Cochran-Mantel-Haenszel — P-value is for overall distribution of responses; Adjusted for baseline lower urinary tract symptoms (LUTS) severity

13. Secondary Outcome: Change in Post Void Residual (PVR) Volume From Baseline to 26 Weeks
Description: Postvoid Residual Volume (PVR) is determined using a portable, calibrated ultrasound device. It consists of the average of a minimum of 3 scans where the residual bladder volume was calculated by averaging the most accurate of the 3 imaging attempts.
Time Frame: Baseline, 26 weeks
Population: All randomized participants who received at least 1 dose of the study drug, had baseline and at least 1 post-baseline PVR measurement.
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 307 | 293
milliliters (mL) | -24.8 (73.08) | -23.1 (66.15)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.157, Wilcoxon Rank-Sum test

14. Secondary Outcome: Change in International Index of Erectile Function (IIEF) Question 3 and 4 Scores From Baseline to 4, 12, and 26 Weeks
Description: IIEF Question 3 asks how often a participant was able to penetrate his partner over the past 4 weeks. Scores range from 0 (did not attempt intercourse) to 5 (almost always or always). IIEF Question 4 asks whether/how often a participant was able to maintain an erection after penetration over the past 4 weeks. Scores range from 0 (did not attempt intercourse) to 5 (almost always or always). Least Squares (LS) Mean values were obtained from a mixed model repeated measures (MMRM) analysis. Model includes treatment, region, visit, baseline IIEF, and visit-by-treatment interaction.
Time Frame: Baseline, 4 weeks, 12 weeks, 26 weeks
Population: All randomized participants who received at least 1 dose of the study drug, had baseline and at least 1 post-baseline IIEF Questions 3 and 4 measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 345 | 350
units on a scale
  Question 3 - 4 weeks | 0.42 (0.09) | -0.32 (0.09)
  Question 3 - 12 weeks | 0.72 (0.09) | 0.04 (0.09)
  Question 3 - 26 weeks | 0.68 (0.10) | -0.07 (0.10)
  Question 4 - 4 weeks | 0.49 (0.09) | -0.21 (0.09)
  Question 4 - 12 weeks | 0.74 (0.09) | 0.13 (0.09)
  Question 4 - 26 weeks | 0.68 (0.10) | 0.06 (0.10)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for Question 3 - 4 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 0.74, 95% CI 2-sided [0.49 to 0.98]
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for Question 3 - 12 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 0.68, 95% CI 2-sided [0.43 to 0.93]
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for Question 3 - 26 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 0.75, 95% CI 2-sided [0.48 to 1.02]
Statistical Analysis 4: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for Question 4 - 4 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 0.71, 95% CI 2-sided [0.46 to 0.95]
Statistical Analysis 5: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for Question 4 - 12 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 0.61, 95% CI 2-sided [0.36 to 0.85]
Statistical Analysis 6: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures Analysis — P-value is for Question 4 - 26 weeks; The Kenward-Roger approximation was used to estimate denominator degrees of freedom; LS Mean Difference = 0.62, 95% CI 2-sided [0.35 to 0.89]

ADVERSE EVENTS:
Arm/Group | Screening-Washout and Placebo Lead-In | Tadalafil | Placebo
Serious Adverse Events (participants affected / at risk) | 1/1070 | 9/345 | 5/350
Other Adverse Events (participants affected / at risk) | 153/1070 | 105/345 | 94/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening-Washout and Placebo Lead-In (N=1070) | Tadalafil (N=345) | Placebo (N=350)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — This event resulted in death.
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening-Washout and Placebo Lead-In (N=1070) | Tadalafil (N=345) | Placebo (N=350)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (3) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 3 (3)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1)
Cheilosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 7 (9) | 8 (11) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 4 (4) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 1 (1) | 0 (0)
Fibrosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 6 (6) | 8 (8) | 8 (11)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 13 (14) | 5 (5) | 3 (3)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Endoscopy upper gastrointestinal tract (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gastric ph decreased (Investigations) | 0 (0) | 4 (4) | 1 (2)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oestradiol increased (Investigations) | 12 (12) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Semen volume decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 15 (16) | 6 (7)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 5 (6)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 2 (3)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (13) | 12 (20) | 12 (15)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Libido decreased (Psychiatric disorders) | 4 (4) | 0 (0) | 4 (4)
Loss of libido (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 5 (5)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 3 (3)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Ejaculation delayed (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ejaculation failure (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 5 (5)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Peyronie's disease (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Testicular mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
Dental operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Toe operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 4 (4) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days